CLINICAL TRIAL: NCT00684411
Title: A Pilot Study of Gleevec (Imatinib Mesylate) in Relapsed/Refractory T Cell Non-Hodgkin's Lymphoma
Brief Title: Gleevec in Relapsed/Refractory T Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Novartis (Industry)
Responsible Party: Principal Investigator, Eric Jacobsen, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-063
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Results first posted 2017-01-05 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2016-11

CONDITIONS: T Cell Non-Hodgkin Lymphoma
Keywords: T NHL; Gleevec; imatinib mesylate
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imatinib mesylate (Experimental): The initial starting dose of imatinib mesylate was 400 mg by mouth once daily but intra-patient dose escalation for patients who did not achieve complete response (CR) was built in upon restaging at weeks 8 and 16. At week 8, patients with partial response (PR) or stable disease (SD) were dose escalated to 600 mg. At week 16, if these patients continued in PR or SD, dose escalated to 800 mg and for patients on 400 mg dose escalated to 600 mg. Patients who experienced disease progression could be dose escalated per MD discretion. Patients were treated as long as receiving clinical benefit and no unacceptable toxicity.
  Interventions: Drug: Imatinib mesylate

INTERVENTIONS:
Drug: Imatinib mesylate
  Other Names: Gleevac

SUMMARY:
The purpose of this research study is to evaluate the overall response rate to imatinib mesylate in participants with relapsed or refractory T cell non-Hodgkin's lymphoma. This drug has been used in chronic myeloid leukemia and information from those other research studies suggests that it may help to treat T cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Objective To evaluate the overall response rate

Secondary Objectives To assess the safety and tolerability To assess the duration of response To assess the progression free survival and overall survival

STATISTICAL DESIGN:

This trial will use a single stage design to differentiate a >/= 25% response rate from a </= 5% rate. If observed data is consistent with the alternative response rate of 25%, imatinib would be deemed clinically interesting and worthy of a larger phase II study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed T NHL, excluding T prolymphocytic leukemia, T lymphoblastic lymphoma, and T/NK large granular lymphocytic leukemia.
* Measurable disease, defined as at least one bidimensionally measurable site of disease measuring at least 1.5cm in greatest diameter.
* Failed at least one systemic chemotherapy or biologic therapy for T cell lymphoma unless it can be clearly documented that the patient can not tolerate such therapy.
* 18 years of age or older
* Life expectancy of greater than 3 months
* ECOG Performance Status of lesser then or equal to 2
* Normal organ and marrow function as outlined in the protocol
* Agree to the use of adequate contraception prior to study entry and for the duration of the study

Exclusion Criteria:

* Chemotherapy or radiotherapy within 4 weeks prior to entering the study
* Receiving any other study agents
* CNS lymphoma requiring active therapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to imatinib mesylate
* Participants requiring concomitant administration of any medications or substances that are inhibitors or inducers of CYP3A4 are ineligible
* Patient previously received radiotherapy to 25% or greater of the bone marrow
* Uncontrolled intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or lactating women
* History of a different malignancy except for individuals who have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy
* HIV-positive individuals on combination antiretroviral therapy
* Known chronic liver disease
* Major surgery within 2 weeks prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jacobsen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jacobsen E, Pozdnyakova O, Redd R, Fisher DC, Dorfman DM, Dal Cin P, LaCasce A, Armand P, Hochberg E, Cote G, Shahsafaei A, Neuberg D, Brown JR, Freedman AS. Imatinib mesylate lacks efficacy in relapsed/refractory peripheral T cell lymphoma. Leuk Lymphoma. 2015 Apr;56(4):993-8. doi: 10.3109/10428194.2014.941835. Epub 2014 Aug 20. PMID 25012943

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 participants were enrolled between August 2008 and December 2011.
Period: Overall Study
Arm/Group | Imatinib Mesylate
Started | 12
Disease Evaluable | 11
Completed | 0
Not Completed | 12
Not completed — New Primary Cancer | 1
Not completed — Disease Progression | 10
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 70.7 [40 to 82]
Gender [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 12
International Prognostic Index (IPI) [Number; unit: participants] — Low risk: 0 - 1 points, low-intermediate risk: 2 points, high-intermediate risk: 3 points, high risk: 4 - 5 points based on risk factors of >60 years of age; stage III or IV disease; elevated serum LDH; ECOG performance status 2, 3 or 4; and >1 extranodal site.
  participants
    Low | 3
    Low-Intermediate | 5
    High-Intermediate | 3
    High | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate is defined as the proportion of patients who achieve complete remission (CR), complete remission/unconfirmed (CRu) or partial remission (PR) based on International Workshop Criteria (IWC) [Cheson, et al. JCO 2007].
  Per the International Working Group response criteria in lymphoma (Cheson 2007) for target lesions assessed by CT: Complete response (CR): nodes that were greater than 15 mm in greatest transverse diameter at baseline shrank to less than 15 mm in greatest transverse diameter and those that were 11-15 mm in greatest transverse diameter but had a short axis diameter greater than 10 mm had a short axis diameter less than 10mm and a transverse diameter that remained less than 15 mm; partial response (PR) was defined as a decrease in the sum of the product of the diameter of target lesions by more than 50% but not fulfilling criteria for CR. Overall response was defined as CR+PR.
  .
Time Frame: Disease was evaluated radiologically at baseline, weeks 8, 16, 24 and every 12 weeks thereafter on treatment. Treatment duration was a median of 56 days (range 5-253 days).
Population: The analysis dataset is comprised of disease evaluable participants. One patient was ineligible based on diagnosis of diffuse large B-cell lymphoma.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 11
proportion of participants | 0.0 [0.0 to 0.238]

2. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) requiring removal from the study or death. Disease progression was assessed per International Workshop Criteria (IWC) [Cheson, et al. JCO 2007].
  Per International Working Group response criteria in lymphoma progressive disease (PD) was defined as the appearance of new lesions; the sum of the product of the diameter (SPD) increasing ≥50% from nadir (smallest value seen during trial) in nodal target lesions overall; or, in any single nodal target lesion, a node with a short axis > 10 mm must increase > 50% in greatest transverse diameter or a node with short axis <10mm must increase by at least 50% to at least 15 mm x 15 mm or have a greatest transverse diameter greater than 15 mm.
Time Frame: Disease was evaluated radiologically at baseline, on treatment at weeks 8, 16, 24 and every 12 weeks thereafter, off treatment for 6 weeks or until death, whichever occurs first. Treatment duration was a median of 56 days (range 5-253 days).
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 11
days | 21 [15 to 28]

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from study entry to death or date last known alive.
Time Frame: Participants were followed long-term for survival for the earlier of 6 weeks from the end of treatment or death. Maximum follow-up was 288 days in this study cohort.
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Imatinib Mesylate
Number analyzed (Participants) | 11
days | 154 [35 to 242]

ADVERSE EVENTS:
Time Frame: Toxicity was evaluated on treatment at weeks 1, 2, every 4 weeks from week 4 until week 28 and then every 12 weeks thereafter starting with week 36.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv3. Other AEs were defined as events with treatment-attribution of possible, probable or definite and grades 1 or 2 per CTCAEv3.
Arm/Group | Imatinib Mesylate
Serious Adverse Events (participants affected / at risk) | 5/12
Other Adverse Events (participants affected / at risk) | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib Mesylate (N=12)
Hemoglobin (Blood and lymphatic system disorders) | 2
Leukocytes (Investigations) | 1
Lymphophenia (Investigations) | 4
Neutrophils (Investigations) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib Mesylate (N=12)
Hemoglobin (Blood and lymphatic system disorders) | 3
Cardiac (Cardiac disorders) | 1
Vision-blurred (Eye disorders) | 1
Vision-flashing lights/floaters (Eye disorders) | 1
Ocular (Eye disorders) | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 1
Fever w/o neutropenia (General disorders) | 1
Edema head and neck (General disorders) | 1
Edema limb (General disorders) | 2
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 1
Leukocytes (Investigations) | 2
Lymphopenia (Investigations) | 1
Neutrophils (Investigations) | 2
Platelets (Investigations) | 4
Alkaline phosphatase (Investigations) | 1
AST, SGOT (Investigations) | 2
Bilirubin (Investigations) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Bicarbonate (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 2
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No